CLINICAL TRIAL: NCT04142164
Title: Computer-based Tutorial and Automated Speech Recognition as Supportive Means to Enhance the Patient Experience and Improve the Efficiency of the Informed Consent Process for Intravitreal Drug Injections
Brief Title: Computer-based Tutorial and Automated Speech Recognition for Intravitreal Drug Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MacInfo
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Age-related Macular Degeneration; Retinal Vein Occlusion; Diabetic Macular Edema
Keywords: Informed Consent Process
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MacInfo presentation (Active Comparator): Patient will get access to an online version of the MacInfo presentation
  Interventions: Other: MacInfo presentation
- Placebo presentation (Placebo Comparator): Patient will get access to an online version of a placebo presentation
  Interventions: Other: Placebo presentation

INTERVENTIONS:
Other: MacInfo presentation — Presentation about intravitreal drug injection
  Arms: MacInfo presentation
Other: Placebo presentation — Placebo presentation
  Arms: Placebo presentation

SUMMARY:
Evaluation if a computer-based tutorial ("MacInfo" tool) improves the patients' knowledge about intravitreal drug injections, associated risks, and the underlying diseases of treatment-naive patients.

DETAILED DESCRIPTION:
Informing the patient an obtaining informed consent is one of the major duties physicians have to perform before beginning a medical treatment. However, patients often experience the informed consent taking as not satisfying. In the past, several approaches were used to try to improve the informed consent taking, such as printed information sheets and multimedia tools.

A novel concept introduced several years ago is the utilization of a multimedia tool including a so-called traffic light system. At our clinic, a computer-based tutorial for informed consent of patients undergoing cataract surgery ("CatInfo" tool) was developed and tested. The patients see and hear a presentation covering the topics of cataract disease, the surgery, and associated risks and complications. After each chapter a graphic representation of a traffic light is shown on the screen. At this page the patient has three choices: if the patient understood everything and wish to continue, the green bar has to be clicked; if there are further questions, the patient clicks the yellow bar; or if the patient wishes to repeat the chapter due to any reason, the patient clicks the red bar.

In previous studies, it was shown that patients who used the CatInfo tool had better knowledge about cataract surgery compared to the ones that saw a placebo video. Furthermore, the overall satisfaction of patients with the CatInfo tool was high (median 9.1 of 10 measured with a visual analogue scale).

Since many cataract patients benefited from using the CatInfo tool, the idea arose to create and test a similar multimedia information tool for patients receiving a drug injection into the vitreous of the eye for treatment of retinal diseases (e.g. patients suffering from neovascular age-related macular degeneration, diabetic macular edema, or retinal venous occlusive disease). Therefore, the "MacInfo" tool was developed as a multidisciplinary project including patients, graphic designers, and ophthalmologists.

Furthermore, it would be helpful for the physician to have a legal valid and written documentation of the informed consent process, serving as proof that the patient was informed correctly about all necessary topics concerning the medical treatment, expected benefits, risks, complications, etc. A novel and technology-driven approach may be the use of Automated Speech Recognition (ASR). ASR records the informed consent discussion, followed by an algorithmic analysis of the conversation, and a subsequent translation of the interaction into a legally valid document.

The aim of this study is to evaluate if the "MacInfo" tool improves the patients' knowledge about intravitreal drug injections, associated risks and the underlying diseases of treatment-naive patients and if ASR is a suitable technology for improving informed consent process documentation in daily routine.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Patients with a need for intravitreal drug administration: wet, age-related macular degeneration (AMD), diabetic macular edema (DME), or retinal venous occlusion
* No previous intravitreal injections
* Willingness and written informed consent to participate in the study

Exclusion Criteria:

* Not literate in German
* Visual acuity of less than 6/60 in the worse eye
* Severe hearing loss
* Inability to use a touch screen device (e.g. severe tremor, etc.)
* Pregnancy - for women in the reproductive age a pregnancy test is required

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of correctly answered questions between study group and control group | 12 months
  Patients are asked to complete a multiple choice questionnaire concerning intravitreal drug injections. Correctly answered questions will be summated. The more points the better the patients' knowledge about intravitreal drug injections.

SECONDARY OUTCOMES:
Usability of the MacInfo tool | 12 months
  By using an visual analogue scale ranging from 0 (worst usability) to 10 (best usability) patients will be asked about their impression concerning usability of the MacInfo tool

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No